CLINICAL TRIAL: NCT02860715
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GX-I7 in Healthy Volunteers
Brief Title: Clinical Trial of GX-I7 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: GX-I7-HV-001
Record Dates: First submitted 2016-06-15; First posted 2016-08-09 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Safety; Pharmacodynamics; Dose-Limiting Toxicity (DLT); Immunogenicity; Pharmacokinetics
MeSH Terms: interventions — efineptakin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort 1 (Experimental): GX-I7 SC 20㎍/㎏ (8 subjects) / Placebo (2 subjects)
  Interventions: Drug: GX-I7; Drug: Placebo
- Cohort 2 (Experimental): GX-I7 SC 60㎍/㎏ (8 subjects) / Placebo (2 subjects)
  Interventions: Drug: GX-I7; Drug: Placebo
- Cohort 3 (Experimental): GX-I7 IM 60㎍/㎏ (8 subjects) / Placebo (2 subjects)
  Interventions: Drug: GX-I7; Drug: Placebo

INTERVENTIONS:
Drug: GX-I7 — Interleukin-7 (IL-7) is T cell growth factor that can be used for treating lymphopenia patients. GX-I7 is a protein drug recombining human IL-7 and hybrid Fc (hyFc). HyFc made by Genexine is composed of hinge-CH2 region of Immunoglobulin D (IgD) and CH2-CH3 region of Immunoglobulin G4 (IgG4). The recombined region is not exposed and each region's characteristics can reduce immunogenicity and improve the efficacy of drug. Consequently, it will be able to treat the patients with lymphopenia in effective ways.
  Other Names: IL-7-hyFc
Drug: Placebo — This is the placebo of GX-I7 described above.
  Other Names: GX-17 vehicle (formulation buffer)

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose study designed to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of GX-I7 in healthy volunteers.

DETAILED DESCRIPTION:
The subjects who are adequately eligible to attend this clinical trial via screening will be hospitalized one day prior to the injection (Day -1), administered a single dose of GX-I7 solution for subcutaneous injection, and then discharged on Day 3. After completing all scheduled tests at the visit 8 (Day 28), safety-related data of each cohort will be evaluated by Independent Safety Monitoring Committee (SMC). Dose escalation will proceed under the principal investigator, medical monitor, and the sponsor's mutual approval, referring to SMC's evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to give informed consent after listening character of the clinical trial
2. Must be 19-45 years of age, inclusive
3. Weight 50-100kg, BMI 18-30kg/m2
4. Subject who is adequately able to attend the study based on medical history and physical exam, no clinically significant abnormality from vital sign and clinical laboratory values
5. No clinical abnormality from ECG test
6. Non-smoker (no smoking or no use of any product containing nicotine least for one month and negative from urine test)

Exclusion Criteria:

1. Suspected or confirmed malignancy, or has malignancy history
2. Any clinically significant acute or chronic medical condition requiring care of a physician, in liver, biliary tract, renal, nervous system (CNS or peripheral). respiratory system, endocrine (diabetes, hyperlipidemia etc), cardiovascular (congestive heart failure, coronary artery disease, myocardial infarction etc), hematology, malignancy, urinary disease, mental disorder, musculoskeletal disorder, immune system (rheumatoid arthritis, lupus etc), otorhinolaryngologic diseases
3. Positive to HBsAg, hepatitis C virus (HCV) Ab and HIV Ab
4. Are considering or scheduled to undergo any surgical or dental procedure during the study
5. Administered other Investigational Product (IP) by attending other clinical study or biological equivalent study within recent 3 months
6. Any Serious adverse drug reaction (SAR) against vaccines or antibiotics, any medical history with serious allergic diseases
7. Positive from urine drug screen or respiratory alcohol screen at medical screening or check-in
8. History of alcohol, drug, or substance abuse in the past 12 months
9. Consumption of alcohol within 48 hours prior to hospitalization
10. Medications with antacid, analgesic, herbal treatment, vitamin, mineral (except maximum 4 grams of acetaminophen) hormone, steroids, insulin, hypoglycemic drug or other hormone substitute within 14 days before administration
11. Planning pregnancy or donation of sperm/disagreeing proper contraception during the study and 3 months following IP administration
12. Do not have veins suitable for cannulation or multiple venipunctures
13. Any other factor that the Investigator thinks will increase subject risk with participation

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2018-06-02 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events including laboratory abnormality after Single Subcutaneous (SC) Injection of GX-I7 | 4 weeks
  Adverse events after injections.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Assessment: Maximum serum concentration (Cmax) | 4 weeks
  PK Parameters to be assessed by single SC administration will be Cmax.
Pharmacokinetic (PK) Assessment: Time to Cmax (Tmax) | 4 weeks
  PK Parameters to be assessed by single SC administration will be Tmax.
Pharmacokinetic (PK) Assessment: apparent terminal half-life (t1/2) | 4 weeks
  PK Parameters to be assessed by single SC administration will be t1/2. t1/2=lnf(2)/λz (λz: invariable for speed of loss obtained from linear regression analysis in logarithmic plot of terminal phase)
Pharmacokinetic (PK) Assessment: Area under the curve from zero to last time of measurable concentration after single administration by trapezoidal rule (AUCt) | 4 weeks
  PK Parameters to be assessed by single SC administration will be AUC (0-inf).
Pharmacokinetic (PK) Assessment: Area under the curve from zero to infinity (AUC(0-inf)) | 4 weeks
  PK Parameters to be assessed by single SC administration will be AUC(0-inf).
Pharmacodynamic (PD) Assessment: Emax of Absolute Lymphocyte Count (ALC) | 8 weeks
  PD parameters will be determined by Emax of ALC, which will be compared with peripheral baseline.
Pharmacodynamic (PD) Assessment: Area Under The Effect-Time Curve Up To Last Quantifiable Effect (AUEClast) of ALC | 8 weeks
  PD parameters will be determined by AUEClast of ALC, which will be compared with peripheral baseline.

OTHER OUTCOMES:
Exploratory PD (PD) assessment: Change of the ratio of immune cells | 4 weeks
  Change of the ratio of immune cells by flow cytometer
Exploratory PD (PD) assessment: T cells in lymphocytes by flow cytometer | 4 weeks
  Cluster of Differentiation 4 (CD4) T and Cluster of differentiation 8 (CD8) T in lymphocytes by flow cytometer

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lee, M.D, Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kang MC, Choi DH, Choi YW, Park SJ, Namkoong H, Park KS, Ahn SS, Surh CD, Yoon SW, Kim DJ, Choi JA, Park Y, Sung YC, Lee SW. Intranasal Introduction of Fc-Fused Interleukin-7 Provides Long-Lasting Prophylaxis against Lethal Influenza Virus Infection. J Virol. 2015 Dec 9;90(5):2273-84. doi: 10.1128/JVI.02768-15. PMID 26656713
- [Background] Seo YB, Im SJ, Namkoong H, Kim SW, Choi YW, Kang MC, Lim HS, Jin HT, Yang SH, Cho ML, Kim YM, Lee SW, Choi YK, Surh CD, Sung YC. Crucial roles of interleukin-7 in the development of T follicular helper cells and in the induction of humoral immunity. J Virol. 2014 Aug;88(16):8998-9009. doi: 10.1128/JVI.00534-14. Epub 2014 Jun 4. PMID 24899182
- [Background] Ahn SS, Jeon BY, Park SJ, Choi DH, Ku SH, Cho SN, Sung YC. Nonlytic Fc-fused IL-7 synergizes with Mtb32 DNA vaccine to enhance antigen-specific T cell responses in a therapeutic model of tuberculosis. Vaccine. 2013 Jun 12;31(27):2884-90. doi: 10.1016/j.vaccine.2013.04.029. Epub 2013 Apr 23. PMID 23624092
- [Background] Martin CE, van Leeuwen EM, Im SJ, Roopenian DC, Sung YC, Surh CD. IL-7/anti-IL-7 mAb complexes augment cytokine potency in mice through association with IgG-Fc and by competition with IL-7R. Blood. 2013 May 30;121(22):4484-92. doi: 10.1182/blood-2012-08-449215. Epub 2013 Apr 22. PMID 23610371
- [Background] Nam HJ, Song MY, Choi DH, Yang SH, Jin HT, Sung YC. Marked enhancement of antigen-specific T-cell responses by IL-7-fused nonlytic, but not lytic, Fc as a genetic adjuvant. Eur J Immunol. 2010 Feb;40(2):351-8. doi: 10.1002/eji.200939271. PMID 19950168
- [Background] Park SH, Song MY, Nam HJ, Im SJ, Sung YC. Codelivery of IL-7 Augments Multigenic HCV DNA Vaccine-induced Antibody as well as Broad T Cell Responses in Cynomolgus Monkeys. Immune Netw. 2010 Dec;10(6):198-205. doi: 10.4110/in.2010.10.6.198. Epub 2010 Dec 31. PMID 21286380
- [Derived] Lee SW, Choi D, Heo M, Shin EC, Park SH, Kim SJ, Oh YK, Lee BH, Yang SH, Sung YC, Lee H. hIL-7-hyFc, A Long-Acting IL-7, Increased Absolute Lymphocyte Count in Healthy Subjects. Clin Transl Sci. 2020 Nov;13(6):1161-1169. doi: 10.1111/cts.12800. Epub 2020 May 20. PMID 32339447